CLINICAL TRIAL: NCT06360601
Title: The Effect of Intravenous Infusion of Labetalol Versus Hydralazine on Cerebral Hemodynamics of Preeclampsia Patients Prospective Randamized Study
Brief Title: Intravenous Labetalol Versus Hydralazine in Preeclampsia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mai Kamal, Lecturer of anaesthesia, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 36264PR589/3/24
Record Dates: First submitted 2024-03-31; First posted 2024-04-11 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-04

CONDITIONS: Preeclampsia Severe
MeSH Terms: interventions — Labetalol; Hydralazine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Labetalol group (Active Comparator)
  Interventions: Drug: Labetalol Injection
- Hydralazine group (Active Comparator)
  Interventions: Drug: HydrALAZINE Injection

INTERVENTIONS:
Drug: Labetalol Injection — Labetalol intravenous infusion 20ml/hr
  Arms: Labetalol group
Drug: HydrALAZINE Injection — Hydralazine intravenous infusion 5mg/hr
  Arms: Hydralazine group

SUMMARY:
We study the effect of intravenous labetalol versus hydralazine in sever preeclampsia patients on cerebral blood flow and neurological outcome

ELIGIBILITY:
Inclusion Criteria:

* patient with clinical diagnosis of sever preeclampsia

Exclusion Criteria:

Patient with history of previous intracranial lesion Patient with history of heart disease/allergy to drug Patient with history of arrhythmia/anticoagulation Any craniotemporal lesion

-

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female as it get pregnant
Enrollment: 40 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-11-20 (Actual); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Cerebral blood flow | Pre intervention-after one hour of intervention
  Mean cerebral blood flow and cerebral perfusion pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta Univeristy hospitals, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes